CLINICAL TRIAL: NCT02327728
Title: Comparison of Different Botulinum Toxin A Injection Patterns in the Treatment of Blepharospasm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: YangHui (Other)
Responsible Party: Sponsor-Investigator, YangHui, MD, PhD, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZOC00173
Record Dates: First submitted 2014-12-18; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Blepharospasm
Keywords: blepharospasm; botulinum A; injection pattern; tear
MeSH Terms: conditions — Blepharospasm; Lacerations | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- medial lower eyelid waived (Experimental): Botulinum toxin A 10U per eye subcutaneous injection at orbicularis oculi
  Interventions: Procedure: Botulinum toxin A injection (4 sites: 10U); Drug: Botulinum toxin A 10U
- full injection pattern (Active Comparator): Botulinum toxin A 12.5U per eye subcutaneous injection at orbicularis oculi
  Interventions: Procedure: Botulinum toxin A injection (5 sites: 12.5U); Drug: Botulinum toxin A 12.5U

INTERVENTIONS:
Procedure: Botulinum toxin A injection (5 sites: 12.5U)
  Arms: full injection pattern
Procedure: Botulinum toxin A injection (4 sites: 10U)
  Arms: medial lower eyelid waived
Drug: Botulinum toxin A 12.5U
  Arms: full injection pattern
Drug: Botulinum toxin A 10U
  Arms: medial lower eyelid waived

SUMMARY:
To evaluate the efficacy of different botulinum toxin A injection patterns in treating benign essential blepharospasm and to compare their influence on condition of eye surface .

DETAILED DESCRIPTION:
The authors performed a prospective double-blinded randomised clinical trial of 60 patients with an established diagnosis of benign essential blepharospasm from February 2013 to December 2015. Patients received a full injection pattern of 5 sites on one eye and a medial lower eyelid waived injection pattern of 4 sites on the other eye randomly. They were surveyed on ocular surface disease index (OSDI), Jankovic rating scale (JRS), blepharospasm disability index (BSDI) prior to injection and 1week, 1month and 3 months after injection. At these time points, closure of the eyelid, tear break up time (BUT), Schirmer test Ｉ, and lower lid tear meniscus height (TMH) were also measured.

ELIGIBILITY:
Inclusion Criteria:

* had a confirmed diagnosis of bilateral BEB
* a minimum of 24-week period since the last injection was required for all patients who had previously received multiple injections of BoNT-A.

Exclusion Criteria:

* blepharospasm of known etiology (caused by medication, injury, etc.)
* history of surgical intervention for BEB (myectomy or neurectomy)
* current ophthalmologic infection
* apraxia of eyelid opening associated with levator palpebrae dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Changes of Jankovic rating scale (JRS) from baseline at 1week, 1month and 3 months | 3 months
Changes of lower lid tear meniscus height (TMH) from baseline at 1week, 1month and 3 months | 3 months

SECONDARY OUTCOMES:
Changes of blepharospasm disability index (BSDI) from baseline at 1week, 1month and 3 months | 3 months
Changes of ocular surface disease index (OSDI) from baseline at 1week, 1month and 3 months | 3 months
Changes of tear break up time (BUT) from baseline at 1week, 1month and 3 months | 3 months
Changes of closure of the eyelid from baseline at 1week, 1month and 3 months | 3 months
Changes of Schirmer test Ｉ from baseline at 1week, 1month and 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hui Yang, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, SunYat-senU
Locations (1):
- Zhongshan Ophthalmic Center, SunYat-senU, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yang H, Lu J, Zhao X, Ding X, Wang Z, Cai X, Luo Y, Lu L. Comparison of Two Botulinum Neurotoxin A Injection Patterns with or without the Medial Lower Eyelid in the Treatment of Blepharospasm. J Ophthalmol. 2016;2016:5957812. doi: 10.1155/2016/5957812. Epub 2016 Jan 14. PMID 26885381